CLINICAL TRIAL: NCT03429764
Title: Comparative Clinical Evaluation of Internal Mattress Sutures vs Continuous Independent Sling Sutures on Interdental Papilla Height and Periodontal Healing in Esthetic Zone: Randomized Clinical Study
Brief Title: Effect of Different Suturing Technique on Height of Interdental Papilla and Periodontal Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rashmiperio
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Gingival Papillary Blunting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CG),CISS (Active Comparator): continuous independent sling sutures (CISS) will be placed with minimum two intact contact points at the surgical site,
  Interventions: Procedure: CISS
- Test group (TG),VIMS (Experimental): internal mattress suture (VIMS) will be placed with minimum two intact contact points at the surgical site,
  Interventions: Procedure: VIMS

INTERVENTIONS:
Procedure: CISS — continuous independent sling sutures will be placed with minimum two intact contact points at the surgical site
  Arms: Control group (CG),CISS
Procedure: VIMS — internal mattress suture will be placed with minimum two intact contact points at the surgical site
  Arms: Test group (TG),VIMS

SUMMARY:
Comparative clinical evaluation of internal mattress sutures vs continuous independent sling sutures on interdental papilla height and periodontal healing in esthetic zone.

To evaluate the effect of internal mattress suturing technique on interdental papilla height and periodontal healing after periodontal surgery in esthetic zone.

To evaluate the effect of continuous independent sling suturing technique on interdental papilla height and periodontal healing after periodontal surgery in esthetic zone.

DETAILED DESCRIPTION:
In the last decade, esthetics has become a major concern in the periodontal therapy. Modern aesthetic dentistry involves not only the restoration of lost teeth, but increasingly the management and reconstruction of the encasing gingiva. Interdental papilla not only acts as a biological barrier in protecting the periodontal structures but also plays a critical role in aesthetics. Numerous risk factors lead to the development of open gingival embrasures or black triangle. These factors include periodontal disease, length of embrasure area, root angulations, interproximal contact position, triangular shape crowns, and consequence of post periodontal surgery.

Interproximal soft tissue craters formation are the consequences of periodontal surgeries like modified widman flap procedures, osseous surgery. Study shows higher percentage of interproximal soft tissue craters in modified widman flap surgery as compared to osseous surgery at six weeks. This creates difficulty for the therapist and patients in performance and plaque control procedures, leading to persistent soft tissue inflammation and black triangle formation.

Primary closure of interdental area is technically more demanding. In periodontal surgery, the most common method of wound closure uses sutures. The primary objectives of suturing are to stabilize and to secure tissues in their desired locations. Therefore choosing an appropriate suturing technique, thread type, thread diameter and surgical needle as well as using proper surgical knot for each thread material are also critical.

Proper management of supracrestal soft tissue flap along with interdental papilla during suturing appears to be of critical importance in ultimate outcome of surgical periodontal pocket management. Wound healing after periodontal flap surgery is achieved through four precisely and highly programmed phases; hemostasis, inflammation, proliferation and remodelling. Wound stability and undisturbed maturation of a fibrin clot adhering to root surface is one of the prerequisite for optimum periodontal regeneration. Wound stability is achieved by close approximation of wound margins for primary intention healing by proper suturing. Wound integrity during the early healing phase rest primarily on the stabilization of the gingival flaps offered by suturing with primary closure of the wound edges inter-proximally while being maintained in maximum passive contact with the root to minimize the intervening blood clot and to prevent wound contamination Mattress sutures are used for greater flap security and control. They permit more precise flap placement, especially when combined with periosteal stabilization. They also allow for good papillary stabilization and placement. These mattress sutures can be internal or external. The internal mattress sutures are used when it is desirable to have the papilla position more upright in the embrasure space. Literature suggests that these sutures may be used in the anterior region when esthetics ideally required that the papilla fill the entire interdental area Continuous independent sling suture are used when multiple teeth are involved, provides greater distribution of forces on the flaps, minimize need for multiple knots, and allow independent placement of buccal and lingual flaps and permits precise flap placement and also secure multiple interproximal papillae of one flap independently of the other flap.

Thus the most suitable suturing technique to achieve healing by primary intention and connective tissue reattachment/ periodontal regeneration and preservation of interdental soft tissue needs to be explored.

Review of the available literature does not reveal studies conducted to evaluate the effect of vertical mattress suture technique and Continuous independent sling suturing techniques on maintaining the height of interdental papilla and periodontal wound healing.

Considering the above mentioned suture technique to be best for primary closure and regeneration as well as maintaining the supracrestal tissue at the desired location, the present study is intended to determine the influence of internal mattress suture and continuous independent sling suture on height of interdental papilla and periodontal healing in the esthetic zone.

MATERIALS AND METHODS

SUBJECT POPULATION

Participants for the study will be selected from Outpatient Department Of Periodontology And Oral Implantology at, Post Graduate Institute of Dental sciences (PGIDS), Rohtak.

STUDY POPULATION AND DESIGN

The study population will consist of minimum of 40 systemically healthy patients aged 18 to 65 years with chronic periodontitis, pocket depth ≥ 5 mm after completed etiological periodontal therapy, requiring open flap debridement in maxillary esthetic zone.

Patients will be randomized in to two groups (minimum 20 each) i.e test and control group.

1. Control group (CG) -continuous independent sling sutures will be placed with minimum two intact contact points at the surgical site.
2. Test group (TG) -- internal mattress suture will be placed with minimum two intact contact points at the surgical site.

All potential participants would be explained the need and design of the study. Only those participant who consented for the study will be included after obtaining written and verbal informed consent.

METHODOLOGY

Patient will be randomly allocated to control and test groups. The study will be conducted as follows-

PRESURGICAL THERAPY

Phase 1 therapy-Oral hygiene instruction, patient education and motivation. Full mouth supragingival and subgingival scaling and root planning with ultrasonic scaler (EMS Piezon 250, Switzerland), hand scaler and curettes (Hu-Friedy) will be completed. Patient will be re-evaluated for periodontal condition after 6 weeks of phase 1 therapy. Sites with probing depth ≥5 mm will be treated with periodontal surgery. Patient with good oral hygiene standard (plaque index score <1 and low level of residual infection (full mouth bleeding score FMBS <20%) will be considered for periodontal surgery.

PERIODONTAL SURGICAL PROCEDURE

After administration of local anaesthesia, open flap debridement will be done on both control group and test group. Test group patients vertical internal mattress suture will be placed and continuous independent sling suture will be placed in control group.

In internal mattress suture, the suture enters the facial tissue just apical to the base of the papilla, runs across the top of alveolar crest, and penetrates the lingual tissue from the inside-out apical to the base of the lingual papilla. The suture passes back through the lingual papilla from the outside-in, 2 to 3 mm coronal to the previous point of suture penetration, and courses back across the alveolar crest exiting through the facial papilla from the inside-out at a point 2 to 3 mm coronal to the initial facial entry point. The facial and lingual papillae are positioned together and the suture is tied on the facial.

In continuous independent sling suture, the suture is passed through the most anterior facial papilla from outside -in just coronal to the mucogingival junction and looped around the lingual of tooth to engage the next facial papilla. The suture does not enter the lingual flap at this time. The suture is looped around each successive tooth, penetrating the facial papilla just coronal to the mucogingival junction.At distal end of flap, the suture is passed through facial tissue and looped back around the lingual of terminal tooth and through the interdental area mesial to the terminal tooth. The suture is then slung around the facial surface of the terminal tooth towards the distal aspect of lingual flap. Wrapping the suture around the terminal tooth in this fashion allows facial flap to be locked in placed and positioned independently of the lingual or palatal flap. The suture is then looped back around the facial surface of terminal tooth. The suture is passed through the interdental area to engage next papilla on the lingual or palatal flap. The lingual flap is sutured in a similar manner as the facial flap. The suture is tied anteriorly where the suture was initially introduced into the facial tissue.

POST OPERATIVE CARE

Patient will be given both verbal and written instructions about post operative care. He/she will be advised:

To take antibiotic Amoxycillin 500mg 8 hourly for 5 days along with Ibuprofen 400 mg 8 hourly for two days.

Sutures will be removed after 1 week.

CLINICAL PARAMETERS

Full mouth indices to be recorded at baseline and follow up.

Probing pocket depth.

Clinical attachment loss.

Bleeding on probing

Site Specific(baseline on the day of surgery) indices

Plaque index (Silness&Loe)

Gingival index (Loe&Silness)

Pocket probing depth

Clinical attachment loss- measured as a distance from cement-enamel junction to the base of pocket.

Bleeding on probing

Location of crest of free gingival margin in respect to CEJ.

Height of interdental papilla

RADIOGRAPHIC PARAMETER

Intraoral periapical radiographs will be taken for diagnostic purpos PPD and CAL will be measured using UNC 15 periodontal probe at six sites (mesiobuccal, distobuccal, mesiolingual, distolingual, and median points at buccal and lingual aspect).

GI, PI will be measured using UNC 15 periodontal probe at four sites(distobuccal, mesiobuccal, facial, lingual gingival margin)

Papillary height will be measured

1. apical aspect of contact point to tip of papilla and
2. from tip of papilla to the mucogingival junction.

The photographs of interdental papilla will be taken and linear measurements as mentioned above will be done on the photographs with the help of Image J software.

Clinical parameters will be recorded at enrolment, baseline, 3 months, and 6 months of periodontal surgery. Interdental papilla height will also be measured at 3 weeks of periodontal surgery. The patients will be reinforced with oral hygiene instructions at every visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with age 18-65 years and who are systemically healthy.
2. Possessing ≥20 natural teeth
3. Patient with chronic periodontitis ( armitage classification)36
4. Pocket depth ≥ 5mm in maxillary esthetic zone
5. Completed etiological periodontal therapy (oral hygiene instructions and scaling and root planning with full-mouth bleeding score FMBS <20% and plaque index score<1 (sillness n loe)37

Exclusion Criteria:

1. Smokers (current and past) and tobacco chewers.
2. Medically compromised patients.
3. Patient on long term use of drugs which could affect the treatment and final outcome of the surgery.
4. Patient under systemic antibiotics in past 6 month.
5. Pregnant women and lactating mothers.
6. Patient who had undergone periodontal treatment 6 months prior to the study.
7. Patients who are allergic to materials or drugs used in study.
8. Patients having loss of contact point in adjacent teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
inerdental papilla height | 6 months
  effect on interdental papilla height,
CAL | 6 months
  Gain in clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: RASHMI SUHAG, Principal Investigator — Post graduate institute of dental science Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India